CLINICAL TRIAL: NCT07130318
Title: Mediterranean Diet in Familial Mediterranean Fever: Is Fatty Liver Affected by Addition of Elliptical Aerobic Exercise
Brief Title: Mediterranean Diet in Familial Mediterranean Fever: Is Fatty Liver Affected by Addition of Aerobic Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-34
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Familial Mediterranean Fever; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Familial Mediterranean Fever; Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): Familial Mediterranean fever (FMF women ) will be collected in this group. the group OF FMF will contain 20 FMF women. the group will follow their colchicine (traditional daily drug therapy for FMF) in addition to Mediterranean diet for six months. also, this group, Group I, will also perform elliptical aerobic exercise (this exercise will be applied for 40 minutes three times weekly and this exercise will be maintained for 6 months)
  Interventions: Behavioral: exercise plus diet restriction
- group number 2 (Active Comparator): Familial Mediterranean fever (FMF women ) will be collected in this group. the group OF FMF will contain 20 FMF women. the group will follow their colchicine (traditional daily drug therapy for FMF) in addition to Mediterranean diet for six months.
  Interventions: Behavioral: diet restriction

INTERVENTIONS:
Behavioral: exercise plus diet restriction — Familial Mediterranean fever (FMF women ) will be collected in this group. the group OF FMF will contain 20 FMF women. the group will follow their colchicine (traditional daily drug therapy for FMF) in addition to Mediterranean diet for six months. also, this group, Group I, will also perform elliptical aerobic exercise (this exercise will be applied for 40 minutes three times weekly and this exercise will be maintained for 6 months)
  Arms: group number 1
Behavioral: diet restriction — Familial Mediterranean fever (FMF women ) will be collected in this group. the group OF FMF will contain 20 FMF women. the group will follow their colchicine (traditional daily drug therapy for FMF) in addition to Mediterranean diet for six months.
  Arms: group number 2

SUMMARY:
Familial Mediterranean fever (FMF) affect liver and causes some dysfunctions including non-alcoholic fatty liver.. still exercise and diet limitation is the treatment for this case

DETAILED DESCRIPTION:
Familial Mediterranean fever (FMF women with fatty liver) will be collected to be cateogarized to group I or group II. Every group OF FMF will contain 20 FMF women. Both groups will follow their colchicine (traditional daily drug therapy for FMF) in addition to Mediterranean diet for six months. Group I will also perform elliptical aerobic exercise (this exercise will be applied for 40 minutes three times weekly and this exercise will be maintained for 6 months)

ELIGIBILITY:
Inclusion Criteria:

* familial Mediterrean fever women
* obese women
* women who have fatty live (non alcoholic type)

Exclusion Criteria:

* cardiac patients
* respiratory disease
* renal disease
* cancer

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-01-08 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
aspartate transaminase | it will be measured after 6 months
  it is a hepatic enzyme

SECONDARY OUTCOMES:
alanine transaminase | it will be measured after 6 months
  it is a hepatic enzyme
body mass index | it will be measured after 6 months
  it will be measured after patient emptying his bowel and bladder
waist circumference | it will be measured after 6 months
  it will be measured at umbilical level
high density lipoprotein | it will be measured after 6 months
  it will be measured in plasma
triglycerides | it will be measured after 6 months
  it will be measured in plasma
cholesterol | it will be measured after 6 months
  it will be measured in plasma
low density lipoprotein | it will be measured after 6 months
  it will be measured in plasma
c reactive protein | it will be measured after 6 months
  it will be measured in plasma
erythrocyte sedimentation rate | it will be measured after 6 months
  it will be measured in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy Cairo university, Dokki, Giza Governorate, Egypt